CLINICAL TRIAL: NCT04489511
Title: A Phase 2a Study of the Safety, Pharmacokinetics and Pharmacodynamics of STG-001 in Subjects With Stargardt Disease (STGD1) Caused by Autosomal Recessive Mutation in ATP Binding Cassette Subfamily A Member 4 (ABCA4) Gene
Brief Title: Study of STG-001 in Subjects With Stargardt Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stargazer Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STG-001-2a
Record Dates: First submitted 2020-07-21; First posted 2020-07-28 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Stargardt Disease-1
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose 1 (Experimental): STG-001 given orally at Dose 1 once a day for 28 days
  Interventions: Drug: STG-001
- Dose 2 (Experimental): STG-001 given orally at Dose 2 once a day for 28 days
  Interventions: Drug: STG-001

INTERVENTIONS:
Drug: STG-001 — Dose 1 or Dose 2 of STG-001 will be administered daily for 28 days to compare safety, pharmacokinetics and pharmacodynamics in Stargardt disease subjects.

SUMMARY:
This is an open-label, multicenter study in subjects with Stargardt disease, comparing 2 doses of STG-001 with regard to safety, pharmacokinetics and pharmacodynamics.

DETAILED DESCRIPTION:
This is an open-label, multicenter, active treatment study in approximately 12 subjects aged 18 to 55 years (inclusive) with STGD1, genotyped with a minimum of two ABCA4 gene mutations. Treatment course of STG-001 at Dose 1 (Cohort 1) or Dose 2 (Cohort 2) testing doses will be administered once daily for 28 days. Cohorts will run in parallel. Subjects will receive their designated dose daily for 28 days and be monitored for safety measures during the dosing period and for an additional 28 days after dosing (through Day 56).

ELIGIBILITY:
Inclusion Criteria:

1. Understand the study procedures and agree to participate by providing written informed consent.
2. STGD1 caused by autosomal recessive mutation in the ABCA4 gene (i.e. at least 2 mutations), confirmed genotypically by a fully accredited certified central genotyping laboratory.
3. 18 to 55 years of age inclusive.
4. Negative pregnancy testing for women of childbearing potential and highly effective double barrier contraception before, during, and for a period after study treatment as described in the clinical protocol.
5. Primary study eye must have at least one well-demarcated area of significantly reduced autofluorescence as imaged by fundus autofluorescence (FAF)
6. In at least one eye and in the same eye:

   1. ETDRS BCVA of less than or equal to 0.4 logMAR (≤68 letters; 20/50 Snellen equivalent) and greater than or equal to 1.3 logMAR (≥19 letters; 20/400 Snellen equivalent); and
   2. Clinical evidence of a macular lesion phenotypically consistent with Stargardt Disease
7. Naïve to investigational treatment for STGD1 with no history of gene therapy, stem cell therapy, surgical implantation of prosthetic retinal chips or intravitreal or sub-retinal injections. History of experimental oral therapy is allowed if it occurred greater than 3 months prior to Screening.
8. Primary study eye must have clear ocular media and adequate pupillary dilation, including no allergy to dilating eyedrops, to permit good quality retinal imaging.
9. In good general health, aside from STGD1, as judged by Investigator.
10. Willing and able to comply with the protocol, including attending assessment visits.

Exclusion Criteria:

1. The subject is an employee of the Sponsor or study site or immediate family member (e.g., spouse, parent, child, sibling) of the Sponsor or study site.
2. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to Day 1 first dose. Herbal supplements and HRT must be discontinued 7 days prior to Day 1 first dose.
3. Presence of any concurrent ocular disease that would affect study outcomes (e.g., severe cataracts; subjects can be enrolled 3 months after successful cataract surgery).
4. Presence of any meaningful retinopathy/maculopathy/atrophy other than as a result of STGD1 in either eye as determined by the Investigator.
5. Has taken non-approved items (supplement containing vitamin A or beta-carotene, liver-based products, or prescription oral retinoid medications) within 30 days of Screening.
6. Use of medications that may interact with Vitamin A metabolism within 60 days of Screening.
7. Participation in an oral interventional study of a vitamin A derivative up to 3 months prior to Screening.
8. The subject had a history of vitamin A deficiency as defined based upon serum values less than 20 mcg/dl (0.7 μmol/L) or clinical signs during slit lamp examination (conjunctival or corneal xerosis; Bitot's spots; corneal ulcers or scarring not due to trauma or other secondary causes).
9. Presence of significant cardiovascular or cerebrovascular disease, including stroke, within 12 months of entry.
10. Has a clinically significant abnormal electrocardiogram (ECG), or has a corrected QT interval (QTc) that is 450 ms or greater.
11. Resting heart rate outside specified limits (< 40/minute, > 100/min) upon repeated measurement.
12. History of diabetes, hepatitis, pancreatitis, cirrhosis, liver failure, uncontrolled thyroid disease or hypervitaminosis A.
13. Any intraocular surgery or thermal laser within 3 months of trial entry. Any prior thermal laser in the macular region.
14. Any major surgical procedure within one month of Screening or planned or anticipated surgery during the study period.
15. Women who are pregnant, nursing, or planning to become pregnant during the study period.
16. Uncontrolled blood pressure outside specified limits (90 mm Hg > Systolic > 140 mm Hg and/or 40 mm Hg > Diastolic > 90 mm Hg) upon repeated measurement.
17. Clinically significant abnormal lab results at Screening, including liver function test (aspartate transaminase, alanine transaminase, bilirubin and alkaline phosphatase) greater than 1.5 x the upper limit of normal (ULN).
18. Actively participating in an investigational therapy study or have received any investigational therapy within 60 days of Screening or 5 half-lives, whichever is longer.
19. Known serious allergies to the fluorescein dye used to measure intraocular pressure, ocular dilating drops, topical ocular anesthetic, components of the STG-001 formulation or any history of anaphylaxis reaction.
20. In the Investigator's assessment, any acute or chronic medical condition, psychiatric condition, physical examination finding or laboratory abnormality that might increase the risk associated with study participation or administration of study treatment or interfere with the interpretation of study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-04-24 (Actual)

PRIMARY OUTCOMES:
Safety events and Tolerability of STG-001 from baseline to 28 days: adverse events | From baseline to 28 days
  Safety and tolerability of 28 days of daily dosing of 2 doses of STG-001 assessed by Incidence and/or clinically significant changes of a combination of ocular and non-ocular adverse events

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of STG-001 maximum plasma concentration (Cmax) at Day 28 | From baseline to 28 days
  Cmax of 2 doses of STG-001 after 28 days of daily dosing of STG-001 assessed by a validated STG-001 assay
Pharmacokinetics (PK) of STG-001 area under the curve (AUC) at Day 28 | From baseline to 28 days
  Exposure to STG-001 as assessed by calculated AUC of 2 doses of STG-001 after 28 days of daily dosing of STG-001
Pharmacodynamics (PD) of STG-001 change in plasma Retinol-Binding Protein 4 (RBP4) at Day 28 | From baseline to 28 days
  Change in Plasma RBP4 levels from baseline to Day 28 with 2 doses of STG-001 after 28 days of daily dosing of STG-001

CONTACTS AND LOCATIONS:
Overall Officials: Prinicpal Investigator, MD, Principal Investigator — Study Site Director
Locations (5):
- United States (5):
  - Associated Retina Consultants, Phoenix, Arizona
  - Vitreo Retinal Associates, P.A., Gainesville, Florida
  - Casey Eye Institute - OHSU, Portland, Oregon
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Retina Foundation of Southwest, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No